CLINICAL TRIAL: NCT02939573
Title: A Randomized Multicenter Study for Isolated Skin Vasculitis
Acronym: ARAMIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Office of Rare Diseases (ORD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VCRC5562; U54AR057319 (NIH)
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Primary Cutaneous Vasculitis; Cutaneous Polyarteritis Nodosa; IgA Vasculitis; Henoch-Schönlein Purpura
MeSH Terms: conditions — IgA Vasculitis | interventions — Colchicine; Dapsone; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stage 1 (Experimental): Eligible patients will be initially randomized (1:1:1) to receive one of the 3 medications under investigation (colchicine 0.6 mg x 2/day; dapsone 150 mg/day; azathioprine 2 mg/kg/day) for 6 months. Endpoint is response to treatment at month 6 (stage 1).
  Interventions: Drug: Colchicine; Drug: Dapsone; Drug: Azathioprine
- Stage 2 (Experimental): If the patient has to discontinue the study drug within the (stage 1) 6 month study period or during the subsequent follow-up period (up to month 12) because of a lack of response (or failure), flare or side effect, he/she will be randomized again to receive one of the remaining two study drugs (stage 2, with a 1:1 randomization ratio, colchicine 0.6 mg x 2/day; dapsone 150 mg/day; azathioprine 2 mg/kg/day) for 6 months. Endpoint in this second stage will again be the response to treatment at 6 months.
  Interventions: Drug: Colchicine; Drug: Dapsone; Drug: Azathioprine

INTERVENTIONS:
Drug: Colchicine — Randomized to colchicine 0.6 mg x 2/day
  Other Names: Colcrys
Drug: Dapsone — Randomized to dapsone 150 mg/day
  Other Names: DDS; Diaminodiphenylsulfone
Drug: Azathioprine — Randomized to azathioprine 2 mg/kg/day
  Other Names: Imuran

SUMMARY:
Multi-center sequential multiple assignment randomized trial comparing the effectiveness of three different standard of care treatment options for patients with isolated skin vasculitis.

DETAILED DESCRIPTION:
Eligible patients will be initially randomized (1:1:1) to receive one of the 3 medications under investigation (colchicine 0.6 mg x 2/day; dapsone 150 mg/day; azathioprine 2 mg/kg/day) for 6 months. Endpoint is response to treatment at month 6 (stage 1).

If the patient has to discontinue the study drug within the 6 month study period or during the subsequent follow-up period (up to month 12) because of a lack of response (or failure), flare or side effect, he/she will be randomized again to receive one of the remaining two study drugs (stage 2, with a 1:1 randomization ratio) for 6 months. Endpoint in this second stage will again be the response to treatment at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary skin vasculitis, not associated with any significant extra-cutaneous involvement that would require specific immunosuppressive therapy. Eligible patients will have a diagnosis of either:

   * Isolated cutaneous small vessel (SV) or medium-sized vessel (MV) vasculitis or cutaneous polyarteritis nodosa (PAN)
   * IgA vasculitis (IgA, formerly Henoch-Schönlein purpura), without active and/or progressing renal involvement (stable glomerular filtration rate (GFR) >60 ml/min; absence of, or mild-and-stable microscopic hematuria without red blood cell casts; absence of, or mild-and-stable proteinuria (<1g/24 hours); not requiring systemic immunosuppressive therapy).

   These conditions, when skin-limited, are all currently treated in similar manners in practice. Mild arthralgias, myalgias, peripheral limb edema, fatigue, weight loss ≤6 lbs or 3 kg within past 3 months, low-grade fever, and mild anemia (Hb ≥ 10 g/dL) will be allowed.
2. The diagnosis of vasculitis must have been confirmed by skin biopsy prior to enrollment (earlier, at diagnosis, and/or just prior to enrollment) that has included an immunofluorescence study (in the case of small vessel vasculitis).
3. Patients must have active cutaneous vasculitis lasting for at least 1 month continuously and/or have had 2 or more flares over the six months preceding enrollment (post-inflammatory lesions such as hyperpigmentation or healing ulceration(s) are not to be considered active vasculitis).
4. Patients must have active / ongoing cutaneous vasculitis lesions at the time of enrollment (post-inflammatory lesions such as hyperpigmentation or healing ulceration(s) are not to be considered active vasculitis).
5. Patients may have a contra-indication to one of the study drug or have been treated prior to enrollment with one of the study medications but failed to respond to it (according to the study definitions of failure and if they have been on the drug at the target dose or higher for 3 months or longer) or had to stop it because of an adverse event. Such patients can be enrolled directly in the second stage of the study and be randomized to receive one of the two other study drugs. The number of such patients enrolled directly in stage 2 will be capped at 10 (10% of the total recruitment target).
6. Patients may have received systemic glucocorticoids for their cutaneous vasculitis before enrollment. For the patients on prednisone at the time of enrollment, prednisone should be stopped within a maximum of 6 weeks after enrollment and initiation of the study drug, following a pre-defined tapering schedule. Patients on long-term, low and stable dose of glucocorticoids (≤5 mg/day prednisone-equivalent) for other conditions (e.g., asthma or adrenal insufficiency) can be enrolled if the likelihood of requiring a dose increase for this other condition is low during the 6 month study period (these patients will remain on that low and stable dose during the study period, with the option to receive one short course of prednisone at higher doses for skin vasculitis flare during the first 3 months of the study period, like any other patients enrolled).
7. Participant age 18 years or greater.

Exclusion Criteria:

1. Presence of significant extra-cutaneous manifestations suggestive of a systemic vasculitis or more diffuse condition. The presence of mild arthralgias, myalgias, peripheral limb edema, fatigue, weight loss ≤6 lbs or 3 kg within past 3 months, low-grade fever, and mild anemia [Hb ≥ 10 g/dL] are not exclusion criteria. Mild and stable microscopic hematuria without RBC casts and/or mild and stable proteinuria (<1g/24 hours) are not exclusion criteria. These latter patients must not require systemic immunosuppressive therapy because of possible renal involvement and their GFR must be >60 ml/min.
2. Known systemic and/or non-skin-isolated vasculitis, such as granulomatosis with polyangiitis, eosinophilic granulomatosis with polyangiitis, cryoglobulinemic vasculitis, systemic polyarteritis nodosa, central nervous system vasculitis and patients with detectable antineutrophil cytoplasmic antibody (ANCA) by immunofluorescence or ELISA.
3. Hypocomplementemic urticarial vasculitis, cryoglobulinemic vasculitis, and other known secondary skin vasculitides such as those secondary to systemic lupus erythematosus, Sjögren syndrome, another auto-immune condition, a cancer, a hematological disorder, an ongoing active infection, or an ongoing medication. Investigators should consider such underlying diagnoses and perform and interpret appropriate laboratory work-up where indicated based on clinical presentation.
4. History of significant intolerance, allergy or serious adverse events to any of the study medications: such patients can be enrolled directly in the second stage of the study and be randomized to receive one of the two other study drugs. The number of patients enrolled directly in stage 2 of the study will be capped at 10 (10%).
5. Patients who have contra-indications to two or three of the study drugs (azathioprine, colchicine, or dapsone), or have been treated prior to enrollment with two or three of the study drugs but failed to respond to them, or had to stop two or three of them because of adverse events.
6. Deficit in glucose-6-phosphate dehydrogenase (G6PD) or history of hemolytic anemia (all patients must be tested for G6PD at the screening visit to assess for their eligibility): such patients can be enrolled directly in the second stage of the study and be randomized to receive one of the two other study drugs (azathioprine or colchicine). The number of patients enrolled directly in stage 2 of the study will be capped at 10 (10%).
7. Low or absent thiopurine methyltransferase (TPMT) activity (if known, not a requirement for study entry): Patients known to have low or absent TPMT can be enrolled directly in the second stage of the study and be randomized to receive one of the two other study drugs (dapsone or colchicine).
8. Evidence of significant hepatic insufficiency or liver function tests > 2 times the upper limit of normal.
9. Evidence of significant renal insufficiency or creatinine clearance < 60 mL/min.
10. Evidence of significant or symptomatic anemia or Hb < 10 g/dL.
11. Comorbid condition that has moderate or high likelihood of requiring intermittent courses of prednisone within the study period, according to the investigator (e.g. chronic obstructive pulmonary disease (COPD), unstable or severe asthma).
12. Active cancer or history of malignancy within the previous 5 years (patient in remission of a cancer >5 years, or with non-metastatic prostate cancer or treated basal or squamous cell carcinoma of the skin can be enrolled).
13. Active uncontrolled or serious infection that may compromise or contra-indicate the use of the study medications.
14. Patient unable to consent.
15. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the study drugs for the treatment of skin vasculitis. | Response to therapy at month 6 of the pooled study stages 1 and 2.
  Compare response to therapies.

SECONDARY OUTCOMES:
Response rates for each of the study drugs | Response evaluated months 3, 6 and 12
  Proportion of patient with complete response and significant response to therapy at months 3, 6 and 12
Physician's global assessment of response | Assessed at months 0, 1, 3, 6, 9, and 12.
  Health-related quality of life as measured using physician's global assessment scale.
Patient's global assessment of response | Assessed at months 0, 1, 3, 6, 9, and 12.
  Health-related quality of life as measured using patient's global assessment scale.
Skindex29 score | Assessed at months 1, 3, 6, 9, and 12.
  Disease activity measured by response to therapy at months 1, 3, 6, and 12
Health-related quality of life | Assessed at months 1, 3, 6, 9, and 12.
  Health-related quality of life as measured using SF-36 and Patient-Reported Outcomes Measurement Information System (PROMIS)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Micheletti, MD, Study Chair — University of Pennsylvania; Christian Pagnoux, MD, MPH, MSc, Study Chair — University of Toronto/Mount Sinai Hospital
Locations (16):
- United States (12):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, Lake Success, New York
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- Canada (3):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - University of Toronto Mount Sinai Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Tohoku Medical and Pharmaceutical University Hospital, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hahn D, Hodson EM, Craig JC. Interventions for preventing and treating kidney disease in IgA vasculitis. Cochrane Database Syst Rev. 2023 Feb 28;2(2):CD005128. doi: 10.1002/14651858.CD005128.pub4. PMID 36853224
- [Derived] Micheletti RG, Pagnoux C, Tamura RN, Grayson PC, McAlear CA, Borchin R, Krischer JP, Merkel PA; Vasculitis Clinical Research Consortium. Protocol for a randomized multicenter study for isolated skin vasculitis (ARAMIS) comparing the efficacy of three drugs: azathioprine, colchicine, and dapsone. Trials. 2020 Apr 28;21(1):362. doi: 10.1186/s13063-020-04285-3. PMID 32345372
- See also: Vasculitis Clinical Research Consoritum — http://www.rarediseasesnetwork.org/vcrc